CLINICAL TRIAL: NCT00070902
Title: The Effects of Positioning and Adjusting on the Z Joint
Brief Title: Using MRI Scans to Evaluate Spinal Manipulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000123-01 (NIH)
Record Dates: First submitted 2003-10-09; First posted 2003-10-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Lower Back Pain
Keywords: Spinal Manipulation; Chiropractic; Zygapophysial Joints
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Procedure: Lumbar side-posture spinal adjusting

SUMMARY:
Lumbar spinal manipulation, or chiropractic adjusting, is thought to separate the surfaces of the spinal joints and thereby relieve lower back pain. This study will use MRI scans to evaluate the spinal joints before and after spinal manipulation.

DETAILED DESCRIPTION:
Zygapophysial joints, better known as facet or "Z" joints, are located on the back (posterior) of the spine on each side of the vertebrae where it overlaps the neighboring vertebrae. Z joints provide stability and allow the spine to bend and twist. Adhesions in the Z joints may develop following hypomobility of vertebrae. These adhesions may be alleviated by separation (gapping) of the Z joints.

Side posture adjusting (spinal manipulation) is thought by many to gap the Z joints, yet no measurable differences of the Z joints before and after spinal manipulation have ever been published. This study will evaluate gapping of the L3/L4, L4/L5, and L5/S1 Z joints by taking measurements directly from MRI scans of the Z joints before and during positioning for a side posture adjustment, and before and after side posture adjusting.

Health volunteers will be randomly assigned to one of four groups: 1) neutral position followed by side posture positioning (trunk rotated to the volunteer's right); 2) neutral position followed by side posture spinal adjusting followed by neutral positioning; 3) neutral position followed by side posture spinal adjusting, followed by side posture positioning; and 4) neutral position followed by neutral position (control group). MRI scans will be taken with the volunteers in the original neutral position and in the final position (either second neutral position or side posture positioning).

ELIGIBILITY:
Inclusion Criteria:

* Student at the National University of Health Sciences
* 185 pounds or less for males and 145 pounds or less for females
* No previous history of lower back pain lasting more than 2 weeks, or no more than three episodes of back pain of brief duration (1 to 2 weeks) in any given year

Exclusion Criteria:

* History of lower back pain
* Presence of disc degeneration, significant osteoarthritis, scoliosis of greater than 20 degrees (Cobb's angle), or other significant pathology seen on x-rays
* Positive findings on orthopedic or neurologic test
* Pregnancy
* Inability of the examining chiropractor to obtain articular releases (audible pop) during lumbar side posture adjustment given at the conclusion of the examination

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64
Dates: Start 2000-06; Study Completion 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D. Cramer, DC, PhD, Principal Investigator — National University of Health Sciences
Locations (1):
- National University of Health Sciences, Lombard, Illinois, United States

REFERENCES:
- [Background] Cramer GD, Gregerson DM, Knudsen JT, Hubbard BB, Ustas LM, Cantu JA. The effects of side-posture positioning and spinal adjusting on the lumbar Z joints: a randomized controlled trial with sixty-four subjects. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2459-66. doi: 10.1097/00007632-200211150-00008. PMID 12435975
- [Background] Cramer GD, Tuck NR Jr, Knudsen JT, Fonda SD, Schliesser JS, Fournier JT, Patel P. Effects of side-posture positioning and side-posture adjusting on the lumbar zygapophysial joints as evaluated by magnetic resonance imaging: a before and after study with randomization. J Manipulative Physiol Ther. 2000 Jul-Aug;23(6):380-94. doi: 10.1067/mmt.2000.108145. PMID 10951308
- See also: National University of Health Sciences — http://www.nuhs.edu